CLINICAL TRIAL: NCT02204956
Title: Extended Care for Smoking Cessation Following Psychiatric Hospitalization
Brief Title: Smoking Cessation Following Psychiatric Hospitalization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01MH104562 (NIH); 1R01MH104562 (NIH)
Record Dates: First submitted 2014-07-28; First posted 2014-07-31 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Nicotine Dependence
Keywords: Smoking cessation; Tobacco use cessation; Psychiatric comorbidity
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sustained Care (Experimental): A 40-minute, in-hospital motivational counseling session about smoking cessation, 8 Interactive Voice Response (IVR) phone calls and/or texts over 90 days, including the possibility of a warm transfer to a telephone tobacco quit line and up to 8-weeks of free transdermal nicotine patches.
  Interventions: Behavioral: Sustained Care
- Usual Care (Active Comparator): A brief 5-10 minute tobacco education session that all hospitalized smokers will receive, delivered by a hospital nurse. During this session, they will be provided with written handouts describing the stages of readiness for change in quitting, self-monitoring of smoking, self-management of smoking situations, relapse prevention, managing stress, other quitting tips and use of nicotine replacement therapy.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Sustained Care — The Sustained Care intervention includes four main components: 1. a 40-minute individual session about quitting smoking during the hospital stay; 2. a 90-day telephone-based and text messaging program that provides support regarding smoking and nicotine patch use; 3. the opportunity, during the automated calls and texts to be transferred to quit smoking resources, including live telephone quit coaching counseling, web and text-based quit coaching resources; and 4. an 8-week supply of nicotine patches, provided at no cost.
  Arms: Sustained Care
Behavioral: Usual Care — Usual Care includes a brief, 5 - 10 minute education session about quitting smoking, delivered by a hospital nurse during the hospital stay. Written handouts to reinforce the educational session will also be provided.
  Arms: Usual Care

SUMMARY:
Smoking rates among individuals with psychiatric disorders are disproportionately higher than the general population. The majority of psychiatric hospitals ban smoking on hospital grounds, thus providing an opportunity for inpatients to experience abstinence. Yet smokers in inpatient psychiatric settings are infrequently provided with referrals for cessation treatment on discharge (< 1 %) and most resume smoking upon discharge. Therefore, the integration of effective cessation interventions within the current mental health treatment system is a public health priority.

The overall objective of this project is to adapt a Sustained Care (SusC) model to smokers with severe mental illness (SMI) engaged in a psychiatric hospitalization and to conduct a randomized, pragmatic effectiveness trial designed to assess the benefit of this adapted SusC intervention in real-world practice. We will test the hypothesis that, among smokers with SMI in inpatient psychiatric treatment (n = 422), SusC will result in significantly greater rates of cotinine-validated, 7-day point prevalence abstinence at 6- and 12-months compared to a group that receives Usual Care (UC) about smoking cessation. Furthermore, we hypothesize that a higher proportion of SusC vs. UC patients will use evidence-based smoking cessation treatment (counseling and pharmacotherapy) in the month after discharge. We will also explore the effect of SusC on health and health care utilization in the 12 months post-discharge (psychiatric symptoms, psychiatric and medical hospital readmissions and emergency room visits) and the effectiveness of SusC on smoking abstinence in patient diagnostic subgroups.

The expected outcome of this project is a demonstration of the effectiveness of a Sustained Care intervention for smoking cessation in individuals with severe mental illness (SMI) following psychiatric hospitalization. Future studies could extend these findings to individuals with SMI receiving outpatient psychiatric treatment or psychotherapy. Overall, this research would have a significant positive public health impact that will move us closer to the long-term goal of dissemination and integration of the Sustained Care model to increase smoking cessation and decrease smoking related morbidity and mortality in people with severe mental illness.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* current smoker (i.e., at least 5 cigarettes/day when not hospitalized)

Exclusion Criteria:

* current diagnosis of dementia
* Mini-Mental State Examination (MMSE: [45]) score < 24
* patient's inability to provide consent for study participation due to his/her inability to demonstrate an understanding of study procedures as contained in the statement of informed consent, after no more than two explanations
* current diagnosis of mental retardation or autistic disorder
* current primary diagnosis of a (non-nicotine) substance use disorder
* no access to a telephone or inability to communicate by telephone
* no planned discharge to institutional setting
* medical contraindication for the use of nicotine replacement therapy (NRT)
* pregnancy, breastfeeding, or plans to become pregnant within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Biochemically verified smoking abstinence via saliva cotinine | 6 months

SECONDARY OUTCOMES:
Proportion of patients who use smoking cessation medication or counseling following discharge | 6 months

OTHER OUTCOMES:
Incremental cost effectiveness | 6 month
Psychiatric symptoms | 6 months
Hospital readmissions, both psychiatric and medical | 6 months
Emergency room visits, both psychiatric and medical | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A. Rigotti, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Seton Shoal Creek Hospital, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brown RA, Minami H, Hecht J, Kahler CW, Price LH, Kjome KL, Bloom EL, Levy DE, Carpenter KM, Smith A, Smits JAJ, Rigotti NA. Sustained Care Smoking Cessation Intervention for Individuals Hospitalized for Psychiatric Disorders: The Helping HAND 3 Randomized Clinical Trial. JAMA Psychiatry. 2021 Aug 1;78(8):839-847. doi: 10.1001/jamapsychiatry.2021.0707. PMID 33950156